CLINICAL TRIAL: NCT00173134
Title: Investigating the Prevalence of Erectile Dysfunction and Erectile Dysfunction Related Quality of Life of Diabetic Men in Taiwan
Brief Title: The Prevalence of Erectile Dysfunction (ED) and ED Related Quality of Life of Diabetic Men
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700404
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-06

CONDITIONS: Diabetes; Erectile Dysfunction
Keywords: diabetes; erectile dysfunction; erectile dysfunction related quality of life
MeSH Terms: conditions — Diabetes Mellitus; Erectile Dysfunction

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Adult diabetic patients aged above 20 attending the diabetic clinic of National Taiwan University Hospital are invited to attend a face to face screening and interview. After obtaining the informed consent, questionnaires including IIEF, DAN-PSS-SEX and erectile dysfunction effect on quality of lie are filled.Personal data, status of diabetes control and complications of diabetes are recorded.The results will be used to investigate the prevalence of erectile dysfunction of diabetic men in Taiwan and erectile dysfunction related quality of life change.

DETAILED DESCRIPTION:
Adult diabetic patients aged above 20 attending the diabetic clinic of National Taiwan University Hospital are invited to attend a face to face screening and interview. After obtaining the informed consent, questionnaires including IIEF, DAN-PSS-SEX and erectile dysfunction effect on quality of lie are filled.Personal data, status of diabetes control and complications of diabetes are recorded.The results will be used to investigate the prevalence of erectile dysfunction of diabetic men in Taiwan and erectile dysfunction related quality of life change.

ELIGIBILITY:
Inclusion Criteria:

diabetic male age above 20

Exclusion Criteria:

men using any form of erectile dysfunction treatment-

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-05; Study Completion 2006-03

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Ping Liu, M.D., Principal Investigator — Department of Urology, National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- Shih-Ping Liu, Taipei, Taiwan